CLINICAL TRIAL: NCT01713569
Title: Feasibility Study: Histological Characterization of Dermal and Subdermal Thermal Coagulation Points in Rhytidectomy Patients After Treatment With the Ulthera® System
Brief Title: Feasibility Study: Histological Characterization After Treatment With the Ulthera® System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow subject enrollment; study to be obtained is no longer required.
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ULT-122
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2013-11

CONDITIONS: Skin Laxity
Keywords: Ulthera® System; Ultherapy™ Treatment; Ulthera, Inc.; Ultrasound treatment for skin tightening
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Subject 1 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 4 MHz, 4.5mm depth transducer at 1.2 Joules and 30 Watts on the Left side versus 0.9 Joules and 30 Watts on the Right side.
  Interventions: Device: Ulthera Treatment
- Subject 2 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 7 MHz, 3.0mm depth transducer at 1.05 Joules and 25 Watts on the Left side versus 0.75 Joules and 25 Watts on the Right side.
  Interventions: Device: Ulthera Treatment
- Subject 3 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 7 MHz, 3.0mm depth transducer at 0.45 Joules and 15 Watts on the Left side versus 0.35 Joules and 14 Watts on the Right side.
  Interventions: Device: Ulthera Treatment
- Subject 4 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 10 MHz, 1.5mm depth transducer at 0.25 Joules and 5 Watts on the Left side versus 0.18 Joules and 5 Watts on the Right side.
  Interventions: Device: Ulthera Treatment
- Subject 5 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 4 MHz, 4.5mm depth transducer at 0.9 Joules and 30 Watts on the Left side versus 7 MHz, 4.5mm 0.9 Joules and 25 Watts on the Right side.
  Interventions: Device: Ulthera Treatment
- Subject 6 (Active Comparator): Ulthera treatment will be administered to both pre-auricular regions using a 7 MHz, 3.0mm transducer at 0.35 and 14 Watts, and a 4 MHz, 4.5mm depth transducer at 0.9 Joules and 30 Watts on the Left side versus a 7 MHz, 3.0mm depth and 4.5mm depth transducer at 2.0 Joules and 40 Watts on the Right side.
  Interventions: Device: Ulthera Treatment

INTERVENTIONS:
Device: Ulthera Treatment — Focused ultrasound energy delivered below the surface of the skin
  Other Names: Ultherapy™

SUMMARY:
Up to 6 subjects will be enrolled. Subjects who have already chosen to have a surgical facelift procedure will be enrolled. Subjects will receive selective Ulthera® ultrasound exposures in the pre-auricular regions. Subject will return for a follow-up visit up to 48 hours post-treatment, on the day of their rhytidectomy. Study images will be obtained pretreatment, immediately post-treatment, and at the follow-up visit.

DETAILED DESCRIPTION:
This study is a prospective, single-center clinical trial. Subjects will be enrolled at the investigator's discretion if they meet inclusion/ exclusion criteria and provide written informed consent. Enrolled subjects will be treated with an assigned transducer based on their order of enrollment. At the study follow-up visit, subjects will undergo resection of the treated tissue for histological analysis prior to their planned rhytidectomy procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 30 to 65 years scheduled for rhytidectomy.
* Subject in good health.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated.
* Willingness and ability to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
* Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at Visit 1 and be willing and able to use an acceptable method of birth control (e.g., barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history: a) Postmenopausal for at least 12 months prior to study; b) Without a uterus and/or both ovaries; or c) A bilateral tubal ligation at least six months prior to study enrollment.

Exclusion Criteria:

* Presence of an active systemic or local skin disease that may affect wound healing.
* Severe solar elastosis.
* Significant scarring in areas to be treated.
* Open wounds or lesions in the area to be treated.
* Severe or cystic acne on the area to be treated.
* Presence of a metal stent or implant in the facial area to be treated.
* Inability to understand the protocol or to give informed consent.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
To determine the depth of focused thermal injury and thermal injury zone dimensions. | 48 hours post-treatment
  Post-treatment, treated tissue will be resected for histological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Sasaki, MD, Principal Investigator — Sasaki Advanced Aesthetic Medical Center
Locations (1):
- Sasaki Advanced Aesthetic Medical Center, Pasadena, California, United States